CLINICAL TRIAL: NCT01916161
Title: The Influence of Information Sources on Knowledge and Anxiety in Inflammatory Bowel Disease Patients
Status: Completed | Type: Observational
Sponsor: National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Christian Selinger, Consultant Gastroenterologist, National Health Service, United Kingdom
Other Study IDs: IBDINFOSOURCE1
Record Dates: First submitted 2013-07-31; First posted 2013-08-05 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Crohn's Disease; Ulcerative Colitis; Anxiety
Keywords: Crohn's disease; ulcerative colitis; anxiety; patient knowledge; information sources
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IBD patients: Ambulatory patients attending IBD clinics at Leeds Teaching Hospitals
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire

SUMMARY:
Inflammatory Bowel Diseases (IBD) are life-long, incurable illnesses that can have a profound effect on the patients quality of life. Disease education is a corner stone of IBD care to enable patients to take up an active role in their disease management. While patient education is enshrined in the IBD standards, actual patient knowledge is often poor.3 Knowledge is not associated with the level of the patient's educational achievement, but member of patient organisations such as Crohn's and Colitis UK (CCUK) have significantly better knowledge than non-members. This may highlight the positive effects of education offered by CCUK, but it is also conceivable that patients with a greater interest in their disease are more like to join organisations like CCUK. Different sources of patient information may therefore influence what level of disease related knowledge a patient achieves.

Apart from high quality clinical information provided by professional organisation (British Society of Gastroenterology, European Crohn's and Colitis Organisation), the National Health Service and charities (CORE, CCUK), there is also a host of unregulated information available. The emerging dominance of the internet for information gathering has provided easy access for patients to a host of websites providing information on IBD. A number of these provide alternative (not evidence based) views, which could have a potentially negative impact on patient's knowledge. Furthermore patients often share their stories on internet forums and it is likely that those stories share are more likely to represent the extreme ends of disease rather than those experienced by the majority. This could potentially cause anxiety in patients with IBD. The quality of information found on the internet varies widely and up to 50% of websites have been judged as poor. The vast majority of patients with IBD have access to the internet and more than half use to search for health related information.7 We have previously also demonstrated that patients with anxiety have better disease related knowledge of IBD.

ELIGIBILITY:
Inclusion Criteria:

patients attending IBD clinics at Leeds Teaching Hospitals

Exclusion Criteria:

* Individuals who are unable to give informed consent.
* Individuals who do not speak English, as the questionanire is selfadministered.
* Individuals under 18 years of age.
* Individuals who are attending Gastroenterology clinics at Leeds General Infirmary and St. James's University Hospital because of a flare up of disease activity of their ulcerative colitis or Crohn's disease.
* Individuals with Crohn's disease who have a stoma (ileostomy), due to practical difficulties in assessing clinical activity in this patient group (it is not actually possible to calculate the HarveyBradshaw index in patients with an ileostomy).
* Individuals who, in the opinion of the investigator, are not suitable to participate in the study.
* Individuals who refuse to give written, informed consent to be involved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ambulatory patients attending IBD clinics at Leeds Teaching Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
CCKNOW | 12 months
  CCKNOW scores according to preferred information source

SECONDARY OUTCOMES:
HADS-A | 12 months
  HADS-A scores according to preferred information source

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, Yorkshire, United Kingdom